CLINICAL TRIAL: NCT04270539
Title: Effects of Short Daytime Nap on Neurocognitive Functioning and Behavior in Chinese Primary School Children
Brief Title: Effect of Nap on Daytime Functioning in Primary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA1807008
Record Dates: First submitted 2020-02-03; First posted 2020-02-17 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Sleep Deprivation
Keywords: primary school children; nap; sleep deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Experimental group (with daytime classroom nap) versus control group (without nap)
Who Masked: Outcomes Assessor
Masking Description: Assessors who are responsible for conducting the cognitive tests are blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (nap) (Experimental): The experimental group will be allowed to take a brief nap daily on school days during the study period.
  Interventions: Behavioral: Nap
- Control Group (no nap) (No Intervention): The control group will not be allowed to take daily nap on school days during the study period.

INTERVENTIONS:
Behavioral: Nap — Participants will be given 20-min nap opportunity in the classroom on a daily basis during school-days.
  Arms: Experimental Group (nap)

SUMMARY:
Previous studies showed that insufficient sleep has a negative impact on children's physical and psychological health. Napping was found to decrease sleepiness and improve daytime functioning in adults and adolescents. The effects of napping on children, however, is unknown. The current study aims to test the effects of short daytime classroom naps on daytime functioning and behaviour in elementary school children.

DETAILED DESCRIPTION:
This study is an interventional study testing the effects of short daytime nap on children's cognitive functioning and daytime behaviour. Primary school children will be randomised to either experimental (nap) or control group (no nap) by class. Measurements include parent-report questionnaires, children's self-report questionnaires, and cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* Children from grade 1, 2, 3, 5, and 6

Exclusion Criteria:

* Children ages 4 or younger, ages 15 or older

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 654 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in objectively measured cognitive performance (sustained attention) | Day 1 (before napping), Day 1 (after napping), two weeks and two months after intervention
  Reaction time (ms) in psychomotor vigilance task
Change in objectively measured cognitive performance (sustained attention) | Day 1 (before napping), Day 1 (after napping), two weeks and two months after intervention
  Lapses defined by reaction time (RT) more than 500ms in psychomotor vigilance task
Change in objectively measured cognitive performance (inhibitory control) | Day 1 (before napping), Day 1 (after napping), two weeks and two months after intervention
  false alarm rate (%) in Go-no go task
Change in objectively measured cognitive performance (inhibitory control) | Day 1 (before napping), Day 1 (after napping), two weeks and two months after intervention
  reaction time (ms) in Go-no go task
Change in objectively measured cognitive performance (working memory) | Day 1 (before napping), Day 1 (after napping), two weeks and two months after intervention
  reaction time (ms) in match to sample task
Change in objectively measured cognitive performance (working memory) | Day 1 (before napping), Day 1 (after napping), two weeks and two months after intervention
  accuracy in match to sample task

SECONDARY OUTCOMES:
Change in daytime sleepiness | Day 1 (before napping), Day 1 (after napping), two weeks and two months after intervention
  Daytime sleepiness as measured by Pediatric Daytime Sleepiness Scale (PDSS). Higher scores suggest more sleepiness.
Change in daytime behaviour (emotional & behavioural problems) | Day 1 (before napping), Day 1 (after napping), two weeks and two months after intervention
  Daytime behaviors as measured by Strengths and Difficulties Questionnaires (SDQ). Higher scores suggest more emotional and behavioural problems.
Change in daytime behaviour (ADHD symptoms) | Day 1 (before napping), Day 1 (after napping), two weeks and two months after intervention
  Strengths and Weakness of Attention-Deficit/ Hyperactivity-symptoms and Normal-behaviors (SWAN). Higher scores suggest more severe ADHD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Shirley X. Li, PhD, DClinPsy, Principal Investigator — The University of Hong Kong
Locations (1):
- Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided